CLINICAL TRIAL: NCT01723774
Title: A Phase II Trial of Neoadjuvant PD 0332991, a Cyclin-Dependent Kinase (Cdk) 4/6 Inhibitor, in Combination With Anastrozole in Women With Clinical Stage 2 or 3 Estrogen Receptor Positive and HER2 Negative Breast Cancer
Brief Title: PD 0332991 and Anastrozole for Stage 2 or 3 Estrogen Receptor Positive and HER2 Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201301106
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Anastrozole; Goserelin; Surgical Procedures, Operative; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: PIK3CA Wild Type Cohort (Experimental): * Tumor biopsy for testing/research at baseline and Cycle 1 Day 15
  * Cycle 0 is 28 days of anastrozole PO daily and, if premenopausal, goserelin SC every 28 days.
  * Cycles 1-5: PD 0332991 combined with anastrozole (and goserelin if premenopausal) is to be (4) 28-day cycles followed by a 5th cycle of 10-12 days duration consisting of daily PD 0332991 and anastrozole (last dose day before surgery)
  * Standard surgery will be performed per institutional standards 2-4 weeks following the completion of Cycle 4 in those who did not receive Cycle 5. In patients who receive Cycle 5, surgery occurs on Day 11, 12, or 13 of Cycle 5.
  * Patients who derived benefit from the therapy have the option of taking PD 0332991 in combination with endocrine therapy for 23 cycles after surgery and adjuvant chemotherapy and radiation if indicated. It should be re-started at least 4 weeks after the completion of chemotherapy and radiation therapy if these treatments were planned.
  Interventions: Drug: PD0332991; Drug: Anastrozole; Drug: Goserelin; Procedure: Surgery (standard of care); Procedure: Tumor biopsy
- Arm 2: PIK3CA Mutant Type Cohort (Experimental): * Tumor biopsy for testing/research at baseline and Cycle 1 Day 15
  * Cycle 0 is 28 days of anastrozole PO daily and, if premenopausal, goserelin SC every 28 days.
  * Cycles 1-5: PD 0332991 combined with anastrozole (and goserelin if premenopausal) is to be (4) 28-day cycles followed by a 5th cycle of 10-12 days duration consisting of daily PD 0332991 and anastrozole (last dose day before surgery)
  * Standard surgery will be performed per institutional standards 2-4 weeks following the completion of Cycle 4 in those who did not receive Cycle 5. In patients who receive Cycle 5, surgery occurs on Day 11, 12, or 13 of Cycle 5.
  * Patients who derived benefit from the therapy have the option of taking PD 0332991 in combination with endocrine therapy for 23 cycles after surgery and adjuvant chemotherapy and radiation if indicated. It should be re-started at least 4 weeks after the completion of chemotherapy and radiation therapy if these treatments were planned.
  Interventions: Drug: PD0332991; Drug: Anastrozole; Drug: Goserelin; Procedure: Surgery (standard of care); Procedure: Tumor biopsy
- Arm 3: Endocrine Resistant Cohort (Experimental): * Tumor biopsy for testing/research at baseline and Cycle 1 Day 15
  * Cycles 1-5: PD 0332991 combined with anastrozole (and goserelin if premenopausal) is to be (4) 28-day cycles followed by a 5th cycle of 10-12 days duration consisting of daily PD 0332991 and anastrozole (last dose day before surgery)
  * Standard surgery will be performed per institutional standards 2-4 weeks following the completion of Cycle 4 in those who did not receive Cycle 5. In patients who receive Cycle 5, surgery occurs on Day 11, 12, or 13 of Cycle 5.
  * Patients who derived benefit from the therapy have the option of taking PD 0332991 in combination with endocrine therapy for 23 cycles after surgery and adjuvant chemotherapy and radiation if indicated. It should be re-started at least 4 weeks after the completion of chemotherapy and radiation therapy if these treatments were planned.
  Interventions: Drug: PD0332991; Drug: Anastrozole; Drug: Goserelin; Procedure: Surgery (standard of care); Procedure: Tumor biopsy

INTERVENTIONS:
Drug: PD0332991
Drug: Anastrozole
  Other Names: Arimidex®
Drug: Goserelin
  Other Names: Zoladex®; Decapeptide I
Procedure: Surgery (standard of care) — -Breast and axillary lymph node surgery
Procedure: Tumor biopsy

SUMMARY:
A Phase II study to investigate the potential utility of PD 0332991 in the treatment of early stage ER+ Human epidermal growth factor receptor 2 (HER2)- breast cancer, to investigate whether the combination of PD 0332991 and anastrozole is able to: 1) improve the pathologic complete response rate when compared to the historical control of single agent aromatase inhibitors, 2) result in fewer patients with on therapy Ki67>10% compared to historical control.

ELIGIBILITY:
Pre-registration PIK3CA Mutant Inclusion

* Clinical T2-T4c, any N, M0 invasive ER+ (Allred Score of 6-8) and HER2 negative (0 or 1+ by IHC or FISH negative for amplification) breast cancer, by AJCC 7th edition clinical staging, with the goal being surgery to completely excise the tumor in the breast and the lymph node. Note: Patients with invasive ER+ (Allred Score of 6-8) HER2- breast cancer or DCIS in the contralateral breast the patient are eligible
* Female ≥18 years of age
* ECOG performance status of 0, 1 or 2
* Life expectancy > 4 months
* Premenopausal, patient must be willing to comply with pregnancy requirements
* Adequate organ and marrow function

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ ULN
  * AST(SGOT)/ and ALT(SGPT) < 2.5 X ULN
  * Creatinine ≤ ULN
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion

* Prior treatment of this cancer including: surgery, radiation, chemotherapy, biotherapy, hormonal therapy, investigational agent prior to study entry
* Receiving any investigational agents
* Prior therapy with any Cdk4 inhibitor
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant/nursing
* Unwilling to employ adequate contraception
* Known HIV-positive on combination antiretroviral therapy
* Evidence of inflammatory cancer
* Known metastatic disease
* Current use of anticoagulation therapy
* Previous excisional biopsy of the breast cancer or sentinel lymph node biopsy
* Any condition that impairs patient's ability to swallow PD 0332991 tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PD 0332991 or other agents used in the study
* Corrected QT interval >470 msec

Registration PIK3CA Mutant Inclusion The criteria below must be met in addition to the pre-registration criteria, except treatment with endocrine therapy for this cancer is allowed prior to registration

* PIK3CA mutant cohort: tumor PIK3CA mutation present
* Premenopausal women, serum estradiol level in postmenopausal range ≤ 7 days prior to registration

Exclusion Criteria below must be met in addition to the pre-registration criteria -Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delavirdine) or inducers (i.e. dexamethasone, glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort)

PIK3CA Wild Type Inclusion

* Clinical T2-T4c, any N, M0 invasive ER+ (Allred Score of 6-8) and HER2 negative (0 or 1+ by IHC or FISH negative for amplification) breast cancer, by AJCC 7th edition clinical staging, with the goal being surgery to completely excise the tumor in the breast and the lymph node. Note: Patients with invasive ER+ (Allred Score of 6-8) HER2- breast cancer or DCIS in the contralateral breast the patient are eligible
* For the PIK3CA wild type cohort: tumor PIK3CA mutation absent. Note that if a patient did not have sufficient research tissue for PIK3CA sequencing at pre-registration or if PIK3CA sequencing result is delayed, she could be registered and enrolled on the PD991 trial without assigning to a particular cohort at the time of enrollment. PIK3CA sequencing will be performed in the future on tumors collected at subsequent time points to assign the treatment cohort or when the PIK3CA sequencing data is available
* For the endocrine resistant cohort: Ki67 > 10% by central testing at Washington University AMP laboratory from a tumor biopsy performed after at least 2 weeks on neoadjuvant endocrine therapy. Note that prior neoadjuvant endocrine therapy could include any endocrine therapy (including aromatase inhibitor, tamoxifen, fulvestrant) alone or in combination, or endocrine therapy in combination with any investigational agent that is not a Cdk 4/6 inhibitor

  *Patients who had a Day 17 Ki67 > 10% from the NCI9170 trial are eligible for the endocrine resistant cohort
* Female >18 years of age
* ECOG performance status of 0, 1 or 2
* Life expectancy > 4 months
* If premenopausal, patient must be willing to comply with pregnancy requirements
* Adequate organ and marrow function:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ ULN
  * AST(SGOT)/ and ALT(SGPT) < 2.5 X ULN
  * Creatinine ≤ ULN
* In premenopausal women, serum estradiol level in postmenopausal range ≤ 7 days prior to registration.
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion

* Prior treatment of this cancer including: Surgery, Radiation therapy, Chemotherapy, Biotherapy, Hormonal therapy, Investigational agent prior to study entry
* Receiving any other investigational agents
* Prior therapy with any Cdk4 inhibitor
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant/nursing
* Unwilling to employ adequate contraception
* Known HIV-positive on combination antiretroviral therapy
* Evidence of inflammatory cancer
* Known metastatic disease
* Current use of anticoagulation therapy
* Previous excisional biopsy of the breast cancer or sentinel lymph node biopsy
* Any condition that impairs patient's ability to swallow PD 0332991 tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PD 0332991 or other agents used in the study
* Corrected QT interval >470 msec
* Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delavirdine) or inducers (i.e. dexamethasone, glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort)

Endocrine Resistant Inclusion

* Clinical T2-T4c at diagnosis or screening, any N, M0 invasive ER+ (Allred Score at least 3 or > 1% ER positivity) and HER2 negative (0 or 1+ by IHC or FISH negative or equivocal) breast cancer, by AJCC 7th edition clinical staging, with the goal being surgery to completely excise the tumor in the breast and the lymph node. Note: Patients with invasive breast cancer that is ER pos, HER2 neg or equivocal or DCIS in the contralateral breast are eligible; multi-focal diseases are not excluded. The dominant lesion will be followed per protocol
* Ki67 > 10% by central testing at Washington University AMP laboratory from a tumor biopsy performed after at least 2 weeks on neoadjuvant endocrine therapy. If Ki67 is > 10% by local testing, the Ki67 slide and H&E slide need to be reviewed by the study pathologist to confirm eligibility (discuss with Study Chair). For patients external to Washington University, please contact the Washington University coordinator by email so that a screening ID# can be assigned prior to shipment of the slides
* Female ≥ 18 years of age
* ECOG performance status of 0, 1 or 2
* Pre- or post-menopausal women are eligible. If premenopausal, patient must be willing to comply with pregnancy requirements and agrees with GnRH agonist therapy for ovarian suppression during the study
* Adequate organ and marrow function:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ ULN
  * AST(SGOT)/ and ALT(SGPT) < 2.5 X ULN
  * Creatinine ≤ ULN
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion

* Prior treatment of this cancer including: Surgery, Radiation, Chemotherapy
* Receiving any other investigational agents
* Prior therapy with Cdk4 inhibitor
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant/nursing
* Unwilling to employ adequate contraception
* Known HIV-positive on combination antiretroviral therapy
* Known metastatic disease
* Current use of anticoagulation therapy
* Previous excisional biopsy of the breast cancer or sentinel lymph node biopsy
* Any condition that impairs patient's ability to swallow PD 0332991 tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PD 0332991 or other agents used in the study
* Corrected QT interval >470 msec
* Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delavirdine) or inducers (i.e. dexamethasone, glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort)

Adjuvant Inclusion

* Derived benefit from PD 0332991 in the neoadjuvant setting in this trial. This includes the 26 patients who achieved complete cell cycle arrest only after the addition of PD 0332991 (C1D1 Ki67 >2.7% and C1D15 Ki67 ≤ 2.7%) from the main study (PIK3CA WT, mutant, or unknown cohorts) as well as any patients who have a Ki67 ≤ 10% on C1D15 biopsy in the endocrine resistant cohort
* ECOG performance status of 0, 1 or 2
* Premenopausal, patient must be willing to comply with pregnancy requirements laid out
* Adequate organ and marrow function

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ ULN
  * AST(SGOT)/ and ALT(SGPT) ≤ 2.5 X ULN
  * Creatinine ≤ ULN
* Underwent surgery of the breast and axilla for curative intent
* At least 4 weeks post completion of adjuvant chemotherapy and radiation therapy if indicated
* Patients who already started on adjuvant hormonal therapy are eligible under the following conditions:

  * For the 26 patients who enrolled in the initial cohorts and derived benefit from neoadjuvant PD 0332991 (C1D1 Ki67 >2.7% and C1D15 Ki67 ≤ 2.7%), adjuvant PD 0332991 should be initiated as soon as possible if adjuvant hormonal therapy has been initiated and the patient has completed radiation if indicated
  * For patients who enrolled in the endocrine resistant cohort and derived benefit from neoadjuvant PD 0332991 (C1D15 Ki67 ≤ 10%), adjuvant PD 0332991 should be initiated within 6 months or sooner after initation of adjuvant hormonal therapy
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion

* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, ssychiatric illness/social situations that would limit compliance with study requirements
* Pregnant/nursing
* Unwilling to employ adequate contraception
* Known HIV-positive on combination antiretroviral therapy. -Known metastatic disease
* Any condition that impairs patient's ability to swallow PD 0332991 tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PD 0332991 or other agents used in the study
* Corrected QT interval >470 msec
* Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delavirdine) or inducers (i.e. dexamethasone, glucocorticoids, progesterone, rifampin, phenobarbital, St. John's wort)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2026-08-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia X Ma, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bagegni N, Thomas S, Liu N, Luo J, Hoog J, Northfelt DW, Goetz MP, Forero A, Bergqvist M, Karen J, Neumuller M, Suh EM, Guo Z, Vij K, Sanati S, Ellis M, Ma CX. Serum thymidine kinase 1 activity as a pharmacodynamic marker of cyclin-dependent kinase 4/6 inhibition in patients with early-stage breast cancer receiving neoadjuvant palbociclib. Breast Cancer Res. 2017 Nov 21;19(1):123. doi: 10.1186/s13058-017-0913-7. PMID 29162134
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjuvant Continuation: Patients who derived benefit from the therapy have the option of taking PD 0332991 in combination with endocrine therapy for 23 cycles after surgery and adjuvant chemotherapy and radiation if indicated. It should be re-started at least 4 weeks after the completion of chemotherapy and radiation therapy if these treatments were planned.
Period: Neoadjuvant
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort | Adjuvant Continuation
Started | 34 | 16 | 34 | 0
Completed | 27 | 12 | 21 | 0
Not Completed | 7 | 4 | 13 | 0
Not completed — Ki67 > 10% | 4 | 0 | 10 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — Disease progression | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0
Not completed — High estradiol | 0 | 1 | 0 | 0
Period: Adjuvant
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort | Adjuvant Continuation
Started | 0 | 0 | 0 | 7
Completed | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort | Total
Number analyzed (Participants) | 34 | 16 | 34 | 84
Age, Continuous [Median (Full Range); unit: years] | 58 [34 to 79] | 55 [34 to 79] | 53 [30 to 76] | 55.5 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 16 | 34 | 84
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 5
  Not Hispanic or Latino | 34 | 15 | 28 | 77
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 6
  White | 30 | 16 | 24 | 70
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 34 | 16 | 34 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Cell Cycle Arrest at Cycle 1 Day 15 (PIK3CA Wild Type Cohort Only)
Description: Complete cell cycle arrest is defined as Ki67 ≤ 2.7% following 2 weeks of neoadjuvant PD 0332991
Time Frame: At cycle 1 day 15 (2 weeks)
Population: Arm 2 and Arm 3 participants were not evaluable for this outcome measure as it is for Arm 1: PIK3CA Wild Type Cohort only. 5 participants in Arm 1 were not evaluable. 1 participant was not evaluable due to insufficient quality of specimen, 1 participant was not evaluable because she withdrew prior to starting treatment, 2 participants were not evaluable because there was no tumor present on biopsy, and 1 participant was not evaluable because she withdrew prior to cycle 1 day 15 biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 29 | 0 | 0
Participants | 23 |  |

2. Primary Outcome: Number of Participants With Complete Cell Cycle Arrest at Cycle 1 Day 15 (Endocrine Resistant Cohort Only)
Description: Complete cell cycle arrest is defined as Ki67 ≤ 2.7% following 2 weeks of neoadjuvant PD 0332991
Time Frame: At cycle 1 day 15 (2 weeks)
Population: Arm 1 and Arm 2 participants were not evaluable for this outcome measure as it is for Arm 3: Endocrine Resistant Cohort only. 1 participant was not evaluable for this outcome measure as the participant did not have any tissue available at the cycle 1 day 15 biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 0 | 0 | 33
Participants |  |  | 19

3. Secondary Outcome: Number of Participants With Complete Cell Cycle Arrest at Cycle 1 Day 15 ( PIK3CA Mutant Type Cohort Only)
Description: Complete cell cycle arrest is defined as Ki67 ≤ 2.7% following 2 weeks of neoadjuvant PD 0332991
Time Frame: At cycle 1 day 15 (2 weeks)
Population: Arm 1 and Arm 3 participants were not evaluable for this outcome measure as it is for Arm 2: PIK3CA Mutant Type Cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 0 | 16 | 0
Participants |  | 16 |

4. Secondary Outcome: Number of Participants With Complete Cell Cycle Arrest
Description: Compare rate of complete cell cycle arrest (defined as Ki67 ≤ 2.7%) arrest between C1D1 and C1D15
Time Frame: Cycle 1 day 1 and cycle 1 day 15 (2 weeks)
Population: PIK3CA Wild Type Cohort - 5 participants not evaluable. 1 due to insufficient quality of specimen, 1 because she withdrew prior to starting treatment, 2 participants because there was no tumor present on biopsy, and 1 because she withdrew prior to cycle 1 day 15 biopsy. Endocrine Resistant Cohort-1 participant because no tissue available at the cycle 1 day 15 biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 29 | 16 | 33
Participants
  Cycle 1 Day 1 complete cell cycle arrest | 8 | 4 | 0
  Cycle 1 Day 15 complete cell cycle arrest | 23 | 16 | 19

5. Secondary Outcome: Clinical Response Rate
Description: * The clinical response rate is the number of patients whose disease meets the WHO criteria of complete or partial response prior to surgery divided by the total number of eligible patients who began combination neoadjuvant treatment.
  * Complete Response (CR) is defined as the disappearance of all known disease based on a comparison between the pre-treatment measurements and the measurements taken at the completion of neo-adjuvant therapy (that is, at the end of cycle 4 neo-adjuvant combination therapy). In addition there is no appearance of new lesions.
  * Partial Response (PR) is defined as a 50% or greater decrease in the product of the bidimensional measurements of the lesion (total tumor size) between the pre-treatment measurements and the measurements taken at the completion of neo-adjuvant therapy (that is, at the end of cycle 4 neo-adjuvant combination therapy). In addition there can be no appearance of new lesions or progression of any lesion.
Time Frame: 16 weeks
Population: 7 participants in Arm 1 were not evaluable for this outcome measure. 3 participants in Arm 2 were not evaluable for this outcome measure. 12 participants in Arm 3 were not evaluable for this outcome measure. Reasons include patient withdrawal (n=4), progressive disease during cycle 1 (n=2), cycle 1 day 15 Ki67 >10% (n=14) high estradiol (n=1), and adverse event (n=1).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 27 | 13 | 22
Participants | 21 | 10 | 16

6. Secondary Outcome: Radiologic Response Rate
Description: * The radiological response rate is the number of patients whose disease meets with WHO criteria for complete or partial response at the evaluation prior to surgery divided by the total number of eligible patients who began combination neo-adjuvant therapy.
  * Complete Response (CR) is defined as the disappearance of all known disease based on a comparison between the pre-treatment measurements and the measurements taken at the completion of neo-adjuvant therapy (that is, at the end of cycle 4 neo-adjuvant combination therapy). In addition there is no appearance of new lesions.
  * Partial Response (PR) is defined as a 50% or greater decrease in the product of the bidimensional measurements of the lesion (total tumor size) between the pre-treatment measurements and the measurements taken at the completion of neo-adjuvant therapy (that is, at the end of cycle 4 neo-adjuvant combination therapy). In addition there can be no appearance of new lesions or progression of any lesion.
Time Frame: At the end of cycle 4 prior to surgery (estimated to be 16 weeks)
Population: Arm 1 PIK3CA Wild Type Cohort: 23 participants not evaluable due to imaging not being performed. Arm 2 PIK3CA Mutant Type Cohort: 9 participants not evaluable due to imaging not being performed. Arm 3 Endocrine Resistant Cohort: 10 participants not evaluable due to imaging not being performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 11 | 7 | 10
Participants | 7 | 3 | 6

7. Secondary Outcome: Safety of PD 0332991 in Combination in Anastrozole as Measured by Frequency and Grade of Related Adverse Events
Description: The maximum grade for each type of adverse event will be recorded for each patient using the NCI-CTCAE v4.0 coding scheme, and frequency tables will be reviewed to determine patterns. Additionally, the relationship (possibly related, probably related, and definitely related) of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: From start of treatment through 30 days after completion of an estimated 4 months of neoadjuvant therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 34 | 16 | 34
Participants
  Grade 1/2 anemia | 4 | 5 | 7
  Grade 1/2 dry eye | 0 | 0 | 1
  Grade 1/2 constipation | 4 | 3 | 1
  Grade 1/2 diarrhea | 4 | 1 | 0
  Grade 1/2 dry mouth | 0 | 0 | 1
  Grade 1/2 dyspepsia | 1 | 1 | 0
  Grade 1/2 flatulence | 1 | 1 | 1
  Grade 1/2 gastroesophageal reflux disease | 0 | 1 | 0
  Grade 1/2 gastrointestinal pain | 0 | 0 | 1
  Grade 1/2 mucositis oral | 9 | 3 | 3
  Grade 1/2 nausea | 8 | 3 | 10
  Grade 1/2 oral pain | 0 | 0 | 1
  Grade 1/2 rectal pain | 1 | 0 | 0
  Grade 1/2 stomatitis | 1 | 0 | 0
  Grade 1/2 vomiting | 0 | 0 | 2
  Grade 1/2 chills | 2 | 1 | 0
  Grade 1/2 edema limbs | 1 | 0 | 0
  Grade 1/2 fatigue | 15 | 8 | 6
  Grade 1/2 fever | 3 | 0 | 1
  Grade 1/2 localized edema | 0 | 1 | 0
  Grade 1/2 pain | 0 | 0 | 1
  Grade 1/2 shingles | 1 | 0 | 0
  Grade 1/2 sinusitis | 1 | 0 | 0
  Grade 1/2 urinary tract infection | 0 | 0 | 1
  Grade 1/2 seroma | 0 | 0 | 1
  Grade 1/2 alanine aminotransferase increased | 1 | 0 | 0
  Grade 3/4 alanine aminotransferase increased | 1 | 1 | 0
  Grade 1/2 aspartate aminotransferase increased | 1 | 0 | 0
  Grade 3/4 aspartate aminotransferase increased | 1 | 0 | 0
  Grade 1/2 lymphocyte count decreased | 3 | 0 | 1
  Grade 1/2 neutrophil count decreased | 14 | 4 | 12
  Grade 3/4 neutrophil count decreased | 7 | 6 | 13
  Grade 1/2 platelet count decreased | 6 | 5 | 3
  Grade 1/2 weight loss | 1 | 0 | 0
  Grade 1/2 white blood cell decreased | 23 | 6 | 11
  Grade 3/4 white blood cell decreased | 0 | 1 | 2
  Grade 1/2 anorexia | 2 | 3 | 1
  Grade 1/2 hypocalcemia | 3 | 0 | 0
  Grade 1/2 hypokalemia | 1 | 0 | 0
  Grade 1/2 hyponatremia | 1 | 0 | 0
  Grade 1/2 arthralgia | 5 | 4 | 0
  Grade 1/2 back pain | 2 | 1 | 0
  Grade 1/2 bone pain | 1 | 0 | 0
  Grade 1/2 myalgia | 2 | 0 | 1
  Grade 1/2 osteoporosis | 0 | 1 | 0
  Grade 1/2 dizziness | 3 | 0 | 0
  Grade 1/2 dysgeusia | 1 | 0 | 0
  Grade 1/2 headache | 5 | 0 | 2
  Grade 1/2 memory impairment | 1 | 0 | 0
  Grade 1/2 peripheral motor neuropathy | 0 | 0 | 1
  Grade 1/2 peripheral sensory neuropathy | 1 | 0 | 0
  Grade 1/2 confusion | 0 | 1 | 0
  Grade 1/2 depression | 2 | 1 | 0
  Grade 1/2 insomnia | 2 | 0 | 1
  Grade 1/2 pelvic pain | 1 | 0 | 0
  Grade 1/2 allergic rhinitis | 1 | 0 | 0
  Grade 1/2 cough | 2 | 0 | 1
  Grade 1/2 dyspnea | 0 | 1 | 2
  Grade 1/2 epistaxis | 1 | 1 | 1
  Grade 1/2 nasal congestion | 1 | 0 | 0
  Grade 1/2 postnasal drip | 1 | 0 | 0
  Grade 1/2 sore throat | 0 | 0 | 1
  Grade 1/2 alopecia | 1 | 4 | 2
  Grade 1/2 dry skin | 2 | 1 | 1
  Grade 1/2 hyperhidrosis | 2 | 2 | 0
  Grade 1/2 papulopustular rash | 1 | 0 | 0
  Grade 1/2 pruritus | 1 | 1 | 0
  Grade 1/2 rash maculo-papular | 1 | 0 | 0
  Grade 3/4 rash maculo-papular | 1 | 0 | 0
  Grade 1/2 fever blister | 1 | 0 | 0
  Grade 1/2 itching | 0 | 0 | 1
  Grade 1/2 hot flashes | 10 | 7 | 3

8. Secondary Outcome: Number of Participants With a PEPI-0 Score
Description: * Preoperative endocrine prognostic index (PEPI) score is derived from four factors assigned a numerical score following neoadjuvant endocrine therapy, including Ki67 expression in the surgical specimen, pathologic tumor size (indicated as "T" below), lymph node status (indicated as "N" below), and estrogen receptor (ER) level (indicated as ER Allred below).
  * PEPI-0 score indicates T1 or T2, N0, Ki67 < 2.7%, ER Allred > 2.
  * It predicts a low risk of recurrence.
Time Frame: At the time of surgery (estimated to be 5 months)
Population: Some participants were not evaluable for this outcome measure due to participant withdrawal and surgery not completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 32 | 14 | 31
Participants | 3 | 2 | 1

9. Secondary Outcome: Change in Ki67 Level of Tumor Specimens
Description: To assess Ki67 level on serially collected tumor specimens
Time Frame: Pre-treatment and cycle 1 day 15
Population: Only participants who had tissue available at the two time points were evaluable for this outcome measure.
Measure: Mean (Full Range); unit: percentage of Ki67 in tumor sample
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 28 | 16 | 33
percentage of Ki67 in tumor sample
  Pre-treatment | 29.75 [3.63 to 74.00] | 19.76 [2.67 to 44.50] | 33.52 [7.48 to 94.25]
  Cycle 1 Day 15: number analyzed (Participants) | 17 | 16 | 33
  Cycle 1 Day 15 | 8.18 [0.00 to 80.00] | 0.51 [0.00 to 1.97] | 15.27 [0.00 to 97.87]

10. Secondary Outcome: Change in Ki67 Level of Tumor Specimens
Description: To assess Ki67 level on serially collected tumor specimens
Time Frame: Cycle 1 day 15 and at time of surgery (approximately 2-4 weeks post completion of cycle 4 - each cycle is 28 days)
Population: Only participants who had tissue available at the two time points were evaluable for this outcome measure.
Measure: Mean (Full Range); unit: percentage of Ki67 in tumor sample
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 19 | 13 | 12
percentage of Ki67 in tumor sample
  Cycle 1 Day 15 | 11.70 [0.00 to 80.00] | 0.51 [0.00 to 1.97] | 0.97 [0.00 to 6.00]
  At time of surgery | 23.00 [1.91 to 75.63] | 8.75 [0.13 to 74.16] | 2.84 [0.00 to 12.00]

11. Secondary Outcome: Number of Participants With Pathologic Complete Response (pCR)
Description: -A pathologic complete response is defined as no histology evidence of invasive tumor cells in the surgical breast specimen and sentinel or axillary lymph nodes.
Time Frame: At the time of surgery (estimated to be 5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort
Number analyzed (Participants) | 34 | 16 | 34
Participants | 0 | 0 | 0

12. Secondary Outcome: Safety Profile of Study Therapy During Adjuvant Therapy as Measured by Frequency and Grade of Adverse Event
Description: as for outcome 7
Time Frame: From start of adjuvant therapy through 30 days after completion of adjuvant therapy (estimated to be 2 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Continuation
Number analyzed (Participants) | 7
Participants
  Grade 1/2 anemia | 1
  Grade 1/2 blurred vision | 1
  Grade 1/2 watering eyes | 1
  Grade 1/2 diarrhea | 1
  Grade 1/2 gastritis | 1
  Grade 1/2 mucositis oral | 1
  Grade 1/2 nausea | 2
  Grade 1/2 vomiting | 1
  Grade 1/2 fatigue | 1
  Grade 1/2 upper respiratory infection | 1
  Grade 1/2 bruising | 1
  Grade 1/2 aspartate aminotransferase increased | 1
  Grade 1/2 lymphocyte count decreased | 3
  Grade 3/4 lymphocyte count decreased | 2
  Grade 1/2 neutrophil count decreased | 2
  Grade 3/4 neutrophil count decreased | 3
  Grade 1/2 platelet count decreased | 1
  Grade 1/2 white blood cell count decreased | 1
  Grade 3/4 white blood cell count decreased | 2
  Grade 1/2 hyperglycemia | 1
  Grade 1/2 arthralgia | 1
  Grade 1/2 alopecia | 2

13. Secondary Outcome: Overall Survival
Time Frame: 5 years
Reporting Status: Not Posted

14. Secondary Outcome: Relapse-free Survival
Time Frame: 5 years
Reporting Status: Not Posted

15. Secondary Outcome: Local Recurrence Rate
Description: Local recurrence is defined as histologic evidence of ductal carcinoma in situ or invasive breast cancer in the ipsilateral breast or chest wall.
Time Frame: 5 years
Reporting Status: Not Posted

16. Secondary Outcome: Regional Recurrence Rate
Description: Regional recurrence is defined as the cytologic or histologic evidence of disease in the ipsilateral internal mammary, ipsilateral supraclavicular, ipsilateral infraclavicular and/or ipsilateral axillary nodes or soft tissue of the ipsilateral axilla.
Time Frame: 5 years
Reporting Status: Not Posted

17. Secondary Outcome: Distant Recurrence Rate
Description: Distant recurrence is defined as the cytologic, histologic, and/or radiographic evidence of disease in the skin, subcutaneous tissue, lymph nodes (other than local or regional metastasis), lung, bone narrow, central nervous system or histologic and/or radiographic evidence of skeletal or liver metastasis.
Time Frame: 5 years
Reporting Status: Not Posted

18. Secondary Outcome: Rate of Second Primary Breast Cancer
Description: Second primary breast cancer is defined histologic evidence of ductal carcinoma in situ or invasive breast cancer in the contralateral breast or chest wall.
Time Frame: 5 years
Reporting Status: Not Posted

19. Secondary Outcome: Rate of Second Primary Cancer (Non-breast)
Description: Second primary cancer (non-breast) is defined as any non-breast second primary cancer other than squamous or basal cell carcinoma of the skin, melanoma in situ, or carcinoma in situ of the cervix is to be reported and should be confirmed histologically whenever possible.
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment until 30 days following the last day of study treatment. Median treatment length of 122.5 days (full range 5-1615 days).
Arm/Group | Arm 1: PIK3CA Wild Type Cohort | Arm 2: PIK3CA Mutant Type Cohort | Arm 3: Endocrine Resistant Cohort | Adjuvant Continuation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/16 | 4/34 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/34 | 1/16 | 1/34 | 1/7
Other Adverse Events (participants affected / at risk) | 34/34 | 16/16 | 34/34 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: PIK3CA Wild Type Cohort (N=34) | Arm 2: PIK3CA Mutant Type Cohort (N=16) | Arm 3: Endocrine Resistant Cohort (N=34) | Adjuvant Continuation (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonitis (Infections and infestations) | 0 | 0 | 1 | 0
Neutrophil count decrease (Investigations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: PIK3CA Wild Type Cohort (N=34) | Arm 2: PIK3CA Mutant Type Cohort (N=16) | Arm 3: Endocrine Resistant Cohort (N=34) | Adjuvant Continuation (N=7)
Anemia (Blood and lymphatic system disorders) | 6 | 5 | 8 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Vision change (Eye disorders) | 1 | 0 | 0 | 0
Watering eyes (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Bleeding gums (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Broken tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 6 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 4 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 10 | 4 | 4 | 1
Nausea (Gastrointestinal disorders) | 11 | 5 | 11 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach cramping (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 5 | 2
Body aches (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 3 | 1 | 2 | 2
Cold symptoms (General disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 3 | 1 | 0 | 0
Fat necrosis (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 18 | 10 | 10 | 1
Fever (General disorders) | 4 | 0 | 1 | 0
Flu like symptoms (General disorders) | 2 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 1 | 0
Nose pain (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 5 | 1 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Shingles (Immune system disorders) | 1 | 0 | 0 | 0
Axilla infection from surgery (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Labia majora cyst (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral yeast infection (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 1
Thrush (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hand wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 2 | 3 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0 | 3 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 3 | 3 | 0
Lymphocyte count decreased (Investigations) | 4 | 0 | 1 | 5
Neutrophil count decreased (Investigations) | 21 | 10 | 25 | 5
Platelet count decreased (Investigations) | 6 | 5 | 5 | 1
Weight loss (Investigations) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 26 | 8 | 14 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 7 | 2 | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 9 | 2 | 6 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Middle ear inflammation (Nervous system disorders) | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 4 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 3 | 2 | 0
Emotional changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 4 | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 1 | 1 | 0
Genital lump (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Vasomotor symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 2 | 2
Armpit pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry fingertips (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 0
Fever blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1
Itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Macular lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodyesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 0
Hot flashes (Vascular disorders) | 13 | 9 | 6 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1
Superficial throbophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatal hernia (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT01723774/Prot_SAP_001.pdf